CLINICAL TRIAL: NCT04278105
Title: Application of High-definition Transcranial Electrical Stimulation in the Upper Extremity Rehabilitation
Brief Title: High-definition Transcranial Electrical Stimulation for Upper Extremity Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); National Cheng Kung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201909051; MOST-108-2321-B-038-002 (Other Grant/Funding Number: Ministry of Science and Technology, R.O.C. (Taiwan))
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Stroke
Keywords: Stroke, Transcranial electrical stimulation, Upper-limb rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HD-tCES & upper extremity rehabilitation (Experimental): The experiment group will receive HD-tCES combined with upper extremity rehabilitation of affected side.
  Interventions: Device: HD-tCES; Other: Upper extremity rehabilitation
- Sham HD-tCES & upper extremity rehabilitation (Sham Comparator): The sham control group will receive sham HD-tCES combined with upper extremity rehabilitation of affected side.
  Interventions: Device: Sham HD-tCES; Other: Upper extremity rehabilitation

INTERVENTIONS:
Device: HD-tCES — The positions of the lesion side primary motor cortex were defined as C3/C4 according to the international 10-20 system of electroencephalograms. HD-tCES will be applied for 20 minutes at an intensity of 1.0 mA direct current stimulation and a specific-added waveform each time, 3 times a week, lasting for 4 weeks.
  Arms: HD-tCES & upper extremity rehabilitation
Device: Sham HD-tCES — The positions of the lesion side primary motor cortex were defined as C3/C4 according to the international 10-20 system of electroencephalograms. Sham HD-tCES will consist of a 5-second ramp up to 1.0 mA direct current stimulation and a specific-added waveform followed immediately by a 5-second ramp down, no current in the middle 19 minutes 40 seconds, and a ramp-up and ramp-down period during the last 10 seconds.
  Arms: Sham HD-tCES & upper extremity rehabilitation
Other: Upper extremity rehabilitation — Upper extremity rehabilitation programs will be selected and graded in accordance with each patient's upper extremity function and specific aims of activities of daily living. Upper extremity rehabilitation will be provided for 30 minutes each time, 3 times a week, lasting for 4 weeks.

SUMMARY:
Transcranial electrical stimulation (tCES) is a non-invasive and safe treatment, which uses a low direct current or alternating current to change the excitability of the cerebral cortex. The tCES has been applied in clinical trials related to rehabilitation research in recent years, and the safety and effectiveness have also been established. However,the existing tCES products effect on the whole brain networks and lack special waveforms. Therefore, we aim to develop a wearable tCES with high definition and special waveforms in this study. This novel stimulation system will result in more precise and focal stimulation of selected brain regions with special waveforms to display better neuromodulation performance. We expect that the novel high-definition tCES (HD-tCES) combined with the upper extremity rehabilitation can shorten the duration of rehabilitative periods, improve stroke patients' activity of daily living, reduce the care burden of patients' family, and subsequently decrease the cost of health care insurance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years.
2. Unilateral cerebral stroke with hemiplegia in Brunnstrom stage III-V.
3. 6 months to 5 years after stroke.
4. Muscular inelasticity (spasticity) 1-3 on the affected upper limb, evaluated by the Modified Ashworth Scale.

Exclusion Criteria:

1. Extremely sensitive to electrical stimulation and cannot tolerate it.
2. Contracture on upper extremities, and limitation in joint range of motion.
3. The muscle tone was severe spasticity,
4. Ossification or inflammation in muscle tissue.
5. A history of cardiopulmonary disease or arrhythmia.
6. With implantable medical electronic devices, like pacemaker.
7. Pressure sores or wounds on the skin of head and upper extremities.
8. Metal implants in the head (neck).
9. Severe cognitive or psychiatric disorders, such as schizophrenia or dissociative identity disorder.
10. A history of seizure or other brain pathology.
11. Brain surgery or severe brain trauma.
12. Drug or alcohol abuse.
13. Malignant neoplasm or rheumatism disorder, like SLE, RA, or AS.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Fugl-Meyer Assessment upper extremity scale (FMA-UE) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 4-week intervention (within 7 days after the last intervention session)
  The FMA-UE assesses motor functioning of upper extremity. Each movement is estimated by a 3-point scale (0-1-2). The total score of the FMA-UE is 66, and a higher score indicates that the patient has better movement ability.

SECONDARY OUTCOMES:
Change from baseline in the Wolf Motor Function Test (WMFT) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 4-week intervention (within 7 days after the last intervention session)
  The WMFT assesses upper extremity motor ability through timed and functional tasks. The items are rated on a 6-point scale (0-1-2-3-4-5). The total score of the WMFT is 75, with higher scores indicating higher functioning levels.
Change from baseline in the Jebsen-Taylor Hand Function Test (JTT) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 4-week intervention (within 7 days after the last intervention session)
  The JTT assesses hand functions commonly used in activities of daily living. The subtests are scored according to time taken to complete the task. Total score is the sum of time taken for each subtest, with shorter times indicating better performance.
Change from baseline in the Modified Ashworth Scale (MAS) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 4-week intervention (within 7 days after the last intervention session)
  The MAS is commonly used in clinical practice for grading spasticity. The MAS is rated on a 6-point scale (0, 1, 1+, 2, 3, 4), and a higher score indicates that the patient has higher muscle tension. The muscles being assessed include shoulder abductor, elbow flexor, elbow extensor, wrist flexor, and finger flexor.
Change from baseline in the Finger to Nose Test after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 4-week intervention (within 7 days after the last intervention session)
  The Finger to Nose Test assesses coordination of upper-extremity movement. The number of complete nose-target movements during a 20-second period will be recorded.
Incidence of treatment-emergent adverse events [safety and tolerability] | Within 10 minutes after each intervention session (a total of 12 sessions, 3 sessions/week, lasting 4 weeks)
  Immediately after each HD-tCES stimulation, the patient will be questioned about eventual side effect.

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital - Taipei Medical University, Taipei

REFERENCES:
- [Derived] Huang YJ, Wang SM, Chen C, Chen CA, Wu CW, Chen JJ, Peng CW, Lin CW, Huang SW, Chen SC. High-Definition Transcranial Direct Current with Electrical Theta Burst on Post-Stroke Motor Rehabilitation: A Pilot Randomized Controlled Trial. Neurorehabil Neural Repair. 2022 Sep;36(9):645-654. doi: 10.1177/15459683221121751. Epub 2022 Sep 1. PMID 36047662
- [Derived] Wang SS, Huang YJ, Chen JJ, Wu CW, Chen CA, Lin CW, Nguyen VT, Peng CW. Designing and pilot testing a novel high-definition transcranial burst electrostimulation device for neurorehabilitation. J Neural Eng. 2021 Sep 17;18(5). doi: 10.1088/1741-2552/ac23be. PMID 34479230